CLINICAL TRIAL: NCT01172158
Title: A Solution for Medical and Legal Problems Arising From Forgotten Ureteral Stents: Reminder Short Message Service (SMS)
Brief Title: SMS Reminder for Forgotten Ureteral Stents
Acronym: sms&FUS
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Dicle University (Other)
Responsible Party: Dicle University, School of Medicine
Other Study IDs: 1-Dicle University
Record Dates: First submitted 2010-06-29; First posted 2010-07-29 (Estimated); Last update posted 2010-07-29 (Estimated); Status verified 2010-07

CONDITIONS: Stents
Keywords: forgotten ureteral stents, SMS Reminder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Forgotten ureteral stents

SUMMARY:
Ureteral stents has become an indispensable instrument for urology practice as a result of widespread use of endourological interventions. Removal of stents could be sometimes neglected by patients or physicians. This omission may lead to legal and medical problems for urologists, health institutions and also for patients. In this study, the investigators offer a computer program providing two sided recall to prevent this nasty complication with sending automatic message by short message service (SMS) to both the patient and the urologist.

DETAILED DESCRIPTION:
In this study, first an institutional subscription agreement was signed between our university and a mobile phone cell company which is supporting SMS sending program. In the second step, by making software plug-in to our hospital's patient follow up program, two programs were integrated. According to this integration, after stent insertion, in case of entering the numerical code corresponding of ''ureteral stent application'' procedure during the stage of epicrisis preparation, the patient follow up system warns the official recording the epicrisis to enter the stent removal time. Patient follow up system transfers this information to SMS sending program. After several weeks of the procedure, if the stent needs to be removed, the software automatically sends a warning message to the patient and the physician. If the patients attends to urology department and undergoes stent removal, the official enters the code of "endoscopic stent removal" to the patient follow-up program. Then the program stops to send warning message.

By the software plug-in to patient follow up program, SMS sending was made mandatory not to forget or skip none of the patients during the epicrisis writing procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had ureteral stent insertion.

Exclusion Criteria:

* Patients who did not want SMS message from us or want to give cell phone number.

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: First an institutional subscription agreement was signed between our university and a mobile phone cell company which is supporting SMS sending program. In the By making software plug-in to our hospital's patient follow up program, two programs were integrated. According to this integration, after stent insertion, in case of entering the numerical code corresponding of ''ureteral stent application'' procedure during the stage of epicrisis preparation, the patient follow up system warns the official recording the epicrisis to enter the stent removal time. Patient follow up system transfers this information to SMS sending program. After several weeks of the procedure, if the stent needs to be removed, the software automatically sends a warning message to the patient and the physician.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2010-05; Primary Completion 2010-10 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
A solution for medical and legal problems arising from forgotten ureteral stents: Reminder Short Message Service (SMS) | five months
  Primary Outcome Measure will be evaluated with;
  1. Number of the patients who admitted for stent removal will be compared with the patients who did not admit. So the effectivity of the SMS sending proram will be evaluated.
  2. The percentage of complication of forgotten ureteral stent will be calculated. And this rate will be compared with the previous rate of same department and the rates reported in the literature.
  3. Patient satisfaction surveys
  4. The time of the patients admitted. The data obtained from this study will be compared with previous data.

SECONDARY OUTCOMES:
SMS Reminder for Forgotten Ureteral Stents | one year
  Secondary, this practice can be prevalent in all hospitals at the our country.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet A Sancaktutar, Asist Prof., Principal Investigator — Department of Urology, Dicle University School of Medicine
Locations (1):
- Dicle University School of Medicine, Diyarbakır, Turkey (Türkiye)